CLINICAL TRIAL: NCT03817242
Title: Comparison of Half-thickness Tragal Cartilage Graft to Temporalis Fascia Graft
Brief Title: Half-thickness Tragal Cartilage Graft vs Temporalis Fascia Graft Tympanoplasty Type I
Acronym: PTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Reading Hospital, Pakistan (Other Government)
Responsible Party: Principal Investigator, Fazal Wahid, Assistant Professor, Lady Reading Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LadyRH
Record Dates: First submitted 2018-12-28; First posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Hearing Loss,Conductive
Keywords: Cartilage; Hearing loss; Tympanoplasty
MeSH Terms: conditions — Hearing Loss, Conductive; Hearing Loss

STUDY DESIGN:
Intervention Model Description: Tympanoplasty I is performed in these patients in Group 1 tragal cartilage graft is used while in group 2 temporalis fascia graft is used
Oversight: Data Monitoring Committee: No

ARMS (2):
- tympanoplasty with tragal cartilage (Active Comparator): Tympanoplasty was performed using tragal cartilage graft
  Interventions: Procedure: Tympanoplasty using tragal cartilage graft
- tympanoplasty with temporalis fascia (Active Comparator): Tympanoplasty was performed using temporalis fascia graft
  Interventions: Procedure: Tympanoplasty using temporalis fascia graft

INTERVENTIONS:
Procedure: Tympanoplasty using tragal cartilage graft — tympanoplasty type I is performed using tragal cartilage in arm 1
  Arms: tympanoplasty with tragal cartilage
Procedure: Tympanoplasty using temporalis fascia graft — tympanoplasty type I is performed using temporalis fascia in arm 2
  Arms: tympanoplasty with temporalis fascia

SUMMARY:
The rationale of this study is to find out the surgical outcome and success rates of tragal cartilage and temporalis fascia, subsequently to develop guide line in light of the results of this study for our department as our institute is going to follow one patient in one bed policy in future. The purpose of this study is to compare the graft success rate of cartilage versus temporalis fascia in tympanoplasty type I in our institute, as no such study has been conducted in our province before.

DETAILED DESCRIPTION:
Tympanic membrane is forming lateral wall of the middle ear cleft which separates middle ear from the external auditory canal. It is made of three layers except in the upper part (Pars Flaccida). The outer layer of TM (Tympanic Membrane) is made of epithelium; middle layer is fibrous tissue, while inner layer is mucosal lining. The thickness of TM measures 0.1 mm, having diameter of 7-10 mm, weighing approximately 14 mg. The function of TM is to assist in hearing and protection of middle ear from infection. Perforation in tympanic membrane is the loss in continuity of TM layers. The causes of TM perforation may be trauma like blast, accident and firearm or infection of the middle ear like acute or chronic suppurative otitis media. It can also be iatrogenic as in case of placement of grommet for glue ear. The purpose of Tympanoplasty is to reconstruct TM perforation and restores sound conducting mechanism. In 1955, Zoellner and Wullstein used different types of graft materials for tympanoplasty. Later Heermann introduced cartilage palisade graft labeled as Simmering Technique. Similarly Goodhill also introduced first cartilage perichondrium composite graft material. Different graft materials can be used to close the TM defect. Some of these materials are temporalis fascia, tragal cartilage, perichondrium and fat. Temporalis fascia and tragal perichondrium had more anatomic proximity, compliance and translucency. The mode of action of these biological graft materials is that it provides support for the membrane remnant to proliferate and heal the defect. The temporalis fascia is thin, translucent and available in sufficient amount; but due to its close resemblance with tympanomeatal flap in color it may be displaced unintentionally during handling. However the reported success rate of temporalis fascia graft in literature varies from 93 to 97%.

On the other hand cartilage is middle ear friendly and survives for comparatively longer time due to the fact that its nourishment is based on diffusion process. Due to rigid nature of cartilage it prevents medialization of the graft to promontory in case of severe eustachian tube dysfunction. Cartilage graft is used in cases of chronically malfunction eustachian tube, adhesive otitis media, recurrent perforation and large TM perforation. But its demerits are its thick nature which hinders sound conduction and it is limited availability. The success rate of the cartilage graft tympanoplasty varies in the literature from 43 - 100%.

Chronic suppurative otitis media is an endemic health problem in our society. The reasons could be probably low literacy level, communities situated far flung from health facilities, lack of specialist service to the public in outreach area and inappropriate treatment of the middle ear infections. Sufficient number of patient suffering from inactive mucosal chronic otitis media with decreased hearing are presenting to otolaryngology unit. Tympanoplasty is the surgery of choice for chronic otitis media inactive mucosal type.

Hypothesis is that cartilage graft tympanoplasty is more successful than temporalis fascia tympanoplasty.

ELIGIBILITY:
Inclusion Criteria:

* All patients of both genders in the age range 16 - 60 years.
* Inactive mucosal COM remained dry for at least one month.
* Conductive hearing loss with minimum air-bone gap (ABG) of 10 Decibel (dB).
* Middle ear is free of disease.

Exclusion Criteria:

* Attic and / or posterior retraction pocket with cholesteatoma.
* Ossicular chain dysfunction and associated otogenic complication.
* Active mucosal COM.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Graft take up | 06 months of follow up
  the graft take rate is determined in both the groups

SECONDARY OUTCOMES:
Objective change in hearing level | 03 months of follow up
  Change in hearing level is objectively assessed by performing pure tone audiometry and that is recorded in decibels on audiogram

OTHER OUTCOMES:
Hearing satisfaction: whispering test | 05 months of follow up
  Individual hearing satisfaction will be assessed subjectively, by whispering test in which whispering sound is offered to the individual and improvement in hearing level is recorded on proforma

CONTACTS AND LOCATIONS:
Overall Officials: Zahid Nazar, Study Director — Lady Reading Hospital, Peshawar, Pakistan
Locations (1):
- Fazali Wahid, Peshawar, Khyberpakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
This data can be share with other researcher through indexed journal
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: UPTO 5 YEARS
Access Criteria: in 6 months and for 5 years